CLINICAL TRIAL: NCT06092775
Title: Prevalence of Subclinical Vertebral Fractures in Rheumatoid Arthritis and Ankylosing Spondylitis in Egyptian Patients and Its Relation to Some Clinical Data
Brief Title: Prevalence of Subclinical Vertebral Fractures in Rheumatoid Arthritis and Ankylosing Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, BASMA ZARIEF NAGEH FAHMY, Resident doctor, Assiut University
Other Study IDs: Vertebral fractures RA ,AS
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Vertebral Fracture
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RA group: DEXA scan X_rays lumber, dorsal spine
  Interventions: Device: DEXA scan,X_ray
- AS group: DEXA scan X_rays lumber, dorsal spine
  Interventions: Device: DEXA scan,X_ray
- Control group: DEXA scan X_rays lumber, dorsal spine
  Interventions: Device: DEXA scan,X_ray

INTERVENTIONS:
Device: DEXA scan,X_ray — DEXA scan detect osteoporosis
  ,X_ray show subclinical vertebral fractures

SUMMARY:
Study of prevalence of subclinical vertebral fractures in Rheumatoid Arthritis and Ankylosing spondylitis

DETAILED DESCRIPTION:
Detection of the prevalence of subclinical vertebral fractures in Rheumatoid Arthritis and Ankylosing spondylitis Study the relation between vertebral fractures and some clinical data like demographics data, disease duration and disease severity

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling ACR/EULAR 2010 rheumatoid arthritis classification criteria.

Patients diagnosed as ankylosing spondylitis according to ASAS criteria (2000). Age (18-50).

Exclusion Criteria:

* Patient with other autoimmune Rheumatic disease other than RA and AS. Infections including hepatitis C or B, HIV, tuberculosis. RA and AS patients with known vertebral fractures. Malignancy, hypogonadism, thyroid problems, chronic kidney disease, Hypoparathyroidism, Type 1 DM.

Pregnancy and breast-feeding.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: RA patients Age from 25 to 45 AS patients age from 25 to 45 Healthy people age from 25 to 45
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of prevalence of subclinical vertebral fractures in RA ,AS and control group | Baseline
  Detection of prevalence of subclinical vertebral fractures in RA, AS and control group

CONTACTS AND LOCATIONS:
Overall Officials: Doaa ABDELHAFEZ, Associte prof, Study Director — Yes; REEM RAMADAN, Dr, Study Director — Yes

REFERENCES:
- [Background] Hu Z, Zhang L, Lin Z, Zhao C, Xu S, Lin H, Zhang J, Li W, Chu Y. Prevalence and risk factors for bone loss in rheumatoid arthritis patients from South China: modeled by three methods. BMC Musculoskelet Disord. 2021 Jun 12;22(1):534. doi: 10.1186/s12891-021-04403-5. PMID 34118911
- [Background] Phuan-Udom R, Lektrakul N, Katchamart W. The association between 10-year fracture risk by FRAX and osteoporotic fractures with disease activity in patients with rheumatoid arthritis. Clin Rheumatol. 2018 Oct;37(10):2603-2610. doi: 10.1007/s10067-018-4218-8. Epub 2018 Jul 23. PMID 30039267
- [Background] Tavassoli S, Rajaei A, Emam MM, Farsad F. Evaluating the Value-Added of the Trabecular Bone Score in Patients with Rheumatoid Arthritis. Arch Iran Med. 2021 Mar 1;24(3):193-198. doi: 10.34172/aim.2021.30. PMID 33878877
- [Background] Raterman HG, Bultink IE, Lems WF. Osteoporosis in patients with rheumatoid arthritis: an update in epidemiology, pathogenesis, and fracture prevention. Expert Opin Pharmacother. 2020 Oct;21(14):1725-1737. doi: 10.1080/14656566.2020.1787381. Epub 2020 Jul 1. PMID 32605401
- [Background] Compston J, Cooper A, Cooper C, Gittoes N, Gregson C, Harvey N, Hope S, Kanis JA, McCloskey EV, Poole KES, Reid DM, Selby P, Thompson F, Thurston A, Vine N; National Osteoporosis Guideline Group (NOGG). UK clinical guideline for the prevention and treatment of osteoporosis. Arch Osteoporos. 2017 Dec;12(1):43. doi: 10.1007/s11657-017-0324-5. Epub 2017 Apr 19. PMID 28425085
- [Background] Tong JJ, Xu SQ, Zong HX, Pan MJ, Teng YZ, Xu JH. Prevalence and risk factors associated with vertebral osteoporotic fractures in patients with rheumatoid arthritis. Clin Rheumatol. 2020 Feb;39(2):357-364. doi: 10.1007/s10067-019-04787-9. Epub 2019 Nov 5. PMID 31691041
- [Background] Navarro-Compan V, Sepriano A, El-Zorkany B, van der Heijde D. Axial spondyloarthritis. Ann Rheum Dis. 2021 Dec;80(12):1511-1521. doi: 10.1136/annrheumdis-2021-221035. Epub 2021 Oct 6. PMID 34615639
- [Background] Bot SD, Caspers M, Van Royen BJ, Toussaint HM, Kingma I. Biomechanical analysis of posture in patients with spinal kyphosis due to ankylosing spondylitis: a pilot study. Rheumatology (Oxford). 1999 May;38(5):441-3. doi: 10.1093/rheumatology/38.5.441. PMID 10371282
- [Background] Westerveld LA, Verlaan JJ, Oner FC. Spinal fractures in patients with ankylosing spinal disorders: a systematic review of the literature on treatment, neurological status and complications. Eur Spine J. 2009 Feb;18(2):145-56. doi: 10.1007/s00586-008-0764-0. Epub 2008 Sep 13. PMID 18791749
- [Background] Zhang M, Li XM, Wang GS, Tao JH, Chen Z, Ma Y, Li XP. The association between ankylosing spondylitis and the risk of any, hip, or vertebral fracture: A meta-analysis. Medicine (Baltimore). 2017 Dec;96(50):e8458. doi: 10.1097/MD.0000000000008458. PMID 29390254
- [Background] Kendler DL, Bauer DC, Davison KS, Dian L, Hanley DA, Harris ST, McClung MR, Miller PD, Schousboe JT, Yuen CK, Lewiecki EM. Vertebral Fractures: Clinical Importance and Management. Am J Med. 2016 Feb;129(2):221.e1-10. doi: 10.1016/j.amjmed.2015.09.020. Epub 2015 Oct 30. PMID 26524708
- [Background] Guanabens N, Olmos JM, Hernandez JL, Cerda D, Hidalgo Calleja C, Martinez Lopez JA, Arboleya L, Aguilar Del Rey FJ, Martinez Pardo S, Ros Vilamajo I, Suris Armangue X, Grados D, Beltran Audera C, Suero-Rosario E, Gomez Gracia I, Salmoral Chamizo A, Martin-Esteve I, Florez H, Naranjo A, Castaneda S, Ojeda Bruno S, Garcia Carazo S, Garcia Vadillo A, Lopez Vives L, Martinez-Ferrer A, Borrell Panos H, Aguado Acin P, Castellanos-Moreira R, Tebe C, Gomez-Vaquero C; OsteoResSer Working Group of the Spanish Society of Rheumatology. Vertebral fractures are increased in rheumatoid arthritis despite recent therapeutic advances: a case-control study. Osteoporos Int. 2021 Jul;32(7):1333-1342. doi: 10.1007/s00198-021-05824-7. Epub 2021 Jan 18. PMID 33459805
- [Background] Schousboe JT. Epidemiology of Vertebral Fractures. J Clin Densitom. 2016 Jan-Mar;19(1):8-22. doi: 10.1016/j.jocd.2015.08.004. Epub 2015 Sep 5. PMID 26349789
- [Background] Tu PH, Liu ZH, Yeap MC, Liu YT, Li YC, Huang YC, Lin TM, Chen CC. Spinal cord injury and spinal fracture in patients with ankylosing spondylitis. BMC Emerg Med. 2022 May 2;22(1):73. doi: 10.1186/s12873-022-00635-3. PMID 35501709
- [Background] Radner H, Neogi T, Smolen JS, Aletaha D. Performance of the 2010 ACR/EULAR classification criteria for rheumatoid arthritis: a systematic literature review. Ann Rheum Dis. 2014 Jan;73(1):114-23. doi: 10.1136/annrheumdis-2013-203284. Epub 2013 Apr 16. PMID 23592710